CLINICAL TRIAL: NCT01888094
Title: SUBclavian Central Venous Catheters Guidance and Examination by UltraSound : a Randomized Controlled Study Versus Landmark Method
Brief Title: SUBclavian Central Venous Catheters Guidance and Examination by UltraSound
Acronym: SUBGEUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0159
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Requiring Subclavian Vein Cannulation; Adult Patients; Patient Covered by French Health Care System
Keywords: Central venous catheter; Complications; Ultrasound; Subclavian vein cannulation; Critical care; Echocardiography; Chest radiographyiography
MeSH Terms: interventions — Restraint, Physical

ARMS (2):
- ultrasound guided for cannulation and examination (Experimental): Prospective, randomized controlled clinical unicentric study, in ICU, Cannulation of the subclavian venous and examination guided with ultrasound
  Interventions: Other: Ultrasound-guided cannulation and examination
- landmark method and examination with chest radiography (Other): Prospective, randomized controlled clinical unicentric study, in ICU, Cannulation of the subclavian venous and examination guided with ultrasound
  Interventions: Other: Ultrasound-guided cannulation and examination

INTERVENTIONS:
Other: Ultrasound-guided cannulation and examination

SUMMARY:
Prospective, randomized controlled clinical unicentric study, in ICU, Cannulation of the subclavian venous and examination guided with ultrasound

DETAILED DESCRIPTION:
One groupe : Ultrasound guided for cannulation and examination of absence ofcomplications One groupe : landmark method and examination with chest radiography

ELIGIBILITY:
Inclusion Criteria:

* adults patients
* requiring subclavian vein cannulation
* patient covered by french health care system

Exclusion Criteria:

* patient refusal
* requiring vein cannulation femoral or jugular
* we see nothing with echocardiography
* children and not adult patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
procedure time between the beginning of procedure ( TO) and when the catheter is controlled ( T4) between strategy catheter cannulation 'standard' and a strategy called "ultrasound all | at day 1

SECONDARY OUTCOMES:
procedure time Tn-Tn (n 0-5) between the two strategies. | at day 1
incidence of occurrence of complications: pneumothorax, hemothorax, bad positioning (outside of the superior vena cava or the right atrium) between the two strategies | at day 1
failure of technology between the two strategies. | at day 1
occurrence of central venous catheter infection. | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Perbet S, Pereira B, Grimaldi F, Duale C, Bazin JE, Constantin JM. Guidance and examination by ultrasound versus landmark and radiographic method for placement of subclavian central venous catheters: study protocol for a randomized controlled trial. Trials. 2014 May 20;15:175. doi: 10.1186/1745-6215-15-175. PMID 24885789